CLINICAL TRIAL: NCT05139680
Title: Real-World Effectiveness of Tafamidis 80 mg or 61 mg on Neurologic Disease Progression in Patients With Mixed-Phenotype Hereditary Transthyretin Amyloid Cardiomyopathy
Brief Title: A Study to Examine the Clinical Effectiveness of Tafamidis in Patients With Mixed Phenotype Hereditary Transthyretin Amyloidosis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461099
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Hereditary Transthyretin Amyloidosis (ATTRv) Cardiomyopathy (CM), Mixed Phenotype
Keywords: transthyretin; amyloidosis; cardiomyopathy; tafamidis; polyneuropathy; progression
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Amyloidosis; Polyneuropathies; Disease Progression | interventions — tafamidis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with mixed phenotype ATTRv-CM: Hereditary ATTR-CM patients presenting with mixed phenotype
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — 80 or 61 milligrams (mg)
  Other Names: Vyndaqel; Vyndamax

SUMMARY:
This study will examine the clinical effectiveness of Tafamidis in patients with Mixed Phenotype Hereditary Transthyretin Amyloidosis using data that already exist in patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at diagnosis
* Diagnosed with ATTRv-CM, mixed phenotype
* Treated with tafamidis (VYNDAQEL 80 mg [four 20-mg tafamidis meglumine capsules] orally once daily or VYNDAMAX 61 mg [one 61-mg tafamidis capsule] orally once daily) for ≥6 months
* Have had ≥1 pre- and ≥2 post-treatment neurologic assessments

Exclusion Criteria:

* History of organ transplant
* Wild-type TTR genotype
* Individuals who are non-ambulatory
* Prior treatment with any disease-modifying therapy (investigational or approved) alone or in combination, except tafamidis, as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily
* Peripheral neuropathy attributed to causes other than ATTR amyloidosis (e.g., diabetes mellitus, B12 deficiency, HIV infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with mixed-phenotype ATTRv-CM who are treated in the Amyloidosis Program at MedStar.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Streicher N, Amass L, Wang R, Stephens JM, LeMasters T, Raina R, Merrill E, Sheikh FH. Real-World Effectiveness of High-Dose Tafamidis on Neurologic Disease Progression in Mixed-Phenotype Variant Transthyretin Amyloid Cardiomyopathy. Cardiol Ther. 2024 Jun;13(2):359-368. doi: 10.1007/s40119-024-00362-9. Epub 2024 Mar 23. PMID 38521883
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants with mixed-phenotype variant transthyretin amyloid cardiomyopathy (ATTRv-CM) who initiated Tafamidis as either VYNDAQEL 80 milligram (mg) or VYNDAMAX 61 mg in a real world setting, were observed retrospectively in this study. Anonymized data was extracted from participant electronic medical records (EMR): MedStar health system in Washington D.C.(08-March-2023 to 19-May-2023).
Groups:
- Tafamidis: Eligible participants with ATTRv-CM who initiated Tafamidis as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally once daily (QD) or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally QD in a real world setting were included in this observational study.
Period: Overall Study
Arm/Group | Tafamidis
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all eligible participants whose data were included and observed in the study.
Groups:
- Tafamidis: Eligible participants with ATTRv-CM who initiated Tafamidis as either VYNDAQEL 80 mg (four 20-mg tafamidis meglumine capsules) orally QD or VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally QD in a real world setting were included in this observational study.
Arm/Group | Tafamidis
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.20 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Neurologic Disease Progression: Number of Participants According to Muscle Weakness Assessment by Neuropathy Impairment Score (NIS) Subscale Score
Description: Neurologic disease progression meant worsening of neurologic function over the time, is assessed by NIS subscale score in this outcome measure. NIS is a composite neurologic impairment score that assesses muscle weakness, sensation, and reflexes by physical exam. NIS subscale for muscle weakness assessment has a score range from 0 (minimum value) to 192 (maximum value). Lower scores indicates normal to mild impairment. Participants were classified as: no change, increase or decrease in NIS subscale scores from pre-treatment baseline period to post-treatment period. Pre-treatment baseline period: at least 6 months and up to 12 months before treatment initiation. Post-treatment period: at least 6 months after treatment initiation with a +/- 3 months window.
Time Frame: Pre-treatment baseline period to post-treatment period (data for specified duration was extracted from medical records and observed retrospectively in this study from 08-Mar-2023 to 19-May-2023)
Population: All eligible participants whose data were included and observed in the study. Here "Number of Participants Analyzed" signifies the number of participants who were evaluable for this outcome measure and had non-missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 7
Participants
  No change in scores | 2
  Increase in scores | 2
  Decrease in scores | 3

2. Primary Outcome: Neurologic Disease Progression: Number of Participants According to Walking Capacity Assessment by Polyneuropathy Disability (PND) Score
Description: Neurologic disease progression meant worsening of neurologic function over the time, is assessed by PND score in this outcome measure. PND is a scoring system to assess participants' walking capacity. It consists of four stages from stage 0 (no impairment) to stage IV (confined to a wheelchair or bedridden). Lower scores indicates normal to mild impairment. Participants were classified as: no change, increase or decrease in PND scores from pre-treatment to post -treatment period. Pre-treatment baseline period: at least 6 months and up to 12 months before treatment initiation. Post-treatment period: at least 6 months after treatment initiation with a +/- 3 months window.
Time Frame: as for outcome 1
Population: All eligible participants whose data were included and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 10
Participants
  No change in scores | 6
  Increase in scores | 1
  Decrease in scores | 3

3. Primary Outcome: Neurologic Disease Progression: Number of Participants According to Muscle Strength Assessment by Medical Research Council (MRC) Scale
Description: Neurologic disease progression meant worsening of neurologic function over the time, is assessed by MRC scale in this outcome measure. MRC assessed muscle strength using a score of 0 (no contraction) to 5 (normal power), to grade the power of a particular muscle group in relation to the movement of a single joint. The higher scores mean a better outcome. Participants were classified as: no change, increase or decrease in MRC scale score from pre-treatment to post-treatment period. Pre-treatment baseline period: at least 6 months and up to 12 months before treatment initiation. Post-treatment period: at least 6 months after treatment initiation with a +/- 3 months window.
Time Frame: as for outcome 1
Population: All eligible participants whose data were included and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 10
Participants
  No change in scores | 8
  Increase in scores | 1
  Decrease in scores | 1

4. Secondary Outcome: Modified Body Mass Index (mBMI)
Description: mBMI was calculated as the product of BMI in kilogram per meter square (kg/m^2) and serum albumin in gram per litre (g/L) to compensate for peripheral edema. Pre-treatment baseline period: at least 6 months and up to 12 months before treatment initiation. Post-treatment period: at least 6 months after treatment initiation with a +/- 3 months window.
Time Frame: Pre-treatment baseline period, post-treatment period (data for specified duration was extracted from medical records and observed retrospectively in this study from 08-Mar-2023 to 19-May-2023)
Population: All eligible participants whose data were included and observed in the study.
Measure: Mean (Standard Deviation); unit: (kg/m^2)*(g/L)
Arm/Group | Tafamidis
Number analyzed (Participants) | 10
(kg/m^2)*(g/L)
  Pre-Treatment | 1001.06 (269.52)
  Post-Treatment | 1070.92 (232.58)

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected for the study.
Description: Due to nature of data in data sources for the study, individual participant data were not retrieved or validated, and it was not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable participant, identifiable reporter, a suspect product, and event) could not be met.
Arm/Group | Tafamidis
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT05139680/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT05139680/SAP_001.pdf